CLINICAL TRIAL: NCT04018807
Title: MVP RCT: Mind and Voice Project Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Quyen Ngo, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00155614; 5K23AA022641-05 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Physical Health; Mental Health; Alcohol; Use, Problem; Interpersonal Violence
MeSH Terms: conditions — Psychological Well-Being; Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource Pamphlet (Other): Participants will receive a pamphlet detailing mental health and social service providers at the local, state, and national level.
  Interventions: Other: Resource pamphlet
- Remote Therapy (Experimental): Participants will receive eight 30-minute remote therapy sessions over the course of twelve weeks.
  Interventions: Behavioral: Remote Therapy

INTERVENTIONS:
Other: Resource pamphlet — The pamphlet will list violence prevention, mental health, and substance abuse services.
  Arms: Resource Pamphlet
Behavioral: Remote Therapy — Remote therapy sessions will include mindfulness exercises and motivational interviewing techniques.
  Arms: Remote Therapy

SUMMARY:
The study seeks to learn more about the health behaviors of young adults. Health behaviors include relationships, physical and mental health, alcohol use, and conflicts with others. The purpose of this study is to improve prevention and intervention programs for young adults.

ELIGIBILITY:
Inclusion Criteria:

* Prior Alcohol Use
* Interpersonal Violence

Exclusion Criteria:

* Person does not understand/speak English
* Prisoner or person being taken into custody/under house arrest
* Person or parent/guardian unable to give consent due to insufficient cognitive orientation due to unknown reasons
* Person unable to give consent due to insufficient cognitive orientation due to drug or alcohol use/ accidental overdose; given pain medications (fails MMSE)
* Person diagnosed with schizophrenia
* Person is actively suicidal or being treated for self-harm (includes overdose with the intent to harm self - not accidental)
* Person being treated for child abuse situation
* Deaf or visually impaired/illiterate/can't speak
* Screened within last month or already in study
* Combative
* Patient died
* Too sick in emergency department to approach (e.g. - never stabilizes, in trauma bay, intubated, on ventilator, or a Level 1 trauma)
* Person has already refused 2 times

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility, as Measured by Number of Sessions Completed | 12 weeks
  At least 80% of session content completed.
Acceptability, as Measured by Client Satisfaction | 12 weeks
  Client satisfaction is measured by the Client Satisfaction Questionnaire Exit-8, an 8 question survey where a high score indicates client satisfaction.
Usability, as Measured by a Modified Systems Usability Scale | 12 weeks
  System usability is measured by an adapted version of the Systems Usability Scale for the platform used.

CONTACTS AND LOCATIONS:
Overall Officials: Quyen Ngo, PhD, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04018807/ICF_000.pdf